CLINICAL TRIAL: NCT05576506
Title: Application of Hyperspectral Imaging Analysis Technology in the Diagnosis of Colorectal Cancer Based on Colonoscopic Biopsy
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2022-SDU-QILU-G003
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Neoplasms; Colorectal Polyp; Colorectal Adenoma; Colorectal SSA
Keywords: Hyperspectral imaging; Artifitial intelligence; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies from the colonic or rectal polyps will be prospectively collected hyperspectral images and conducted for histology examination and model validation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deep learning algorithm group: After the patient has passed the screening, a routine colonoscopy will be performed, and the target tissue with suspected inflammation or neoplasia will be biopsied. The clinical investigators use the hyperspectral microscope to collect image information of the biopsy tissue in the endoscopy room. After collecting information, biopsy specimens will be routinely processed and sent for pathological diagnosis.

SUMMARY:
The purpose of this study is to develop and validate a deep learning algorithm for the diagnosis of colorectal cancer other colorectal disease by marking and analyzing the characteristics of hyperspectral images based on the pathological results of colonoscopic biopsy, so as to improve the objectiveness and intelligence of early colorectal cancer diagnosis.

DETAILED DESCRIPTION:
Prospectively collect the hyperspectral image information of ordinary colonoscopic biopsy tissue. The colonoscopic biopsy tissue is from the Endoscopy Center of Qilu Hospital of Shandong University. The hyperspectral images are marked based on the biopsy pathological results, and the deep convolutional neural network (DCNN) model is used. With training and verification, develop the Hyperspectral Imaging Artificial Intelligence Diagnostic System (HSIAIDS) .A portion of colonoscopic biopsy tissue will be collected as a prospective test set to prospectively test the diagnostic performance of the HSIAIDS algorithm.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-75 years who undergo the colonoscopy examination and biopsy

Exclusion Criteria:

* patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in colonoscopy
* patients with previous surgical procedures on the gastrointestinal tract.
* patients with contraindications to biopsy
* patients who refuse to sign the informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 18-75 years who undergo the colonoscopy examination and biopsy;
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of HSI artificial intelligence model to identify colorectal adenoma and cancer | 1 year
  Accuracy of hyperspectral imaging (HSI) artificial intelligence model to identify colorectal hyperplastic polyp, adenoma, SSL and colorectal cancer. Accuracy of artificial intelligence models Accuracy = (true positives + true negatives) / total number of subjects * 100%
Sensitivity | 1 year
  Sensitivity of HSI artificial intelligence model Sensitivity = number of true positives / (number of true positives + number of false negatives) * 100%.
Specificity | 1 year
  Specificity of HSI Artificial Intelligence Model Specificity = number of true negatives / (number of true negatives + number of false positives))*100%
Negative predictive values(NPV) | 1 year
  Negative predictive values for HSI artificial intelligence model = number of true negatives / (number of true negatives + number of false negatives)*100%
AUC (95% CI) | 1 year
  area under the receiver operating characteristic curve (AUC)

SECONDARY OUTCOMES:
To record and evaluate any unknown risks and adverse events of hyperspectral imaging in specimen image acquisition | 1 year
  To record and evaluate any unknown risks and adverse events of hyperspectral imaging in specimen image acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Study Chair — Study Principal investigator
Locations (1):
- Qilu hosipital, Jinan, Shandong, China